CLINICAL TRIAL: NCT01606644
Title: Hyperbaric Oxygen - a New Treatment Modality in Patients With Radiation Damaged Salivary Gland Tissue.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lone Forner (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Sponsor-Investigator, Lone Forner, DDS, PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HBO Copenhagen study
Record Dates: First submitted 2010-05-06; First posted 2012-05-28 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Late Effect of Radiation
Keywords: radiation sequelae; hyperbaric oxygen
MeSH Terms: interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HBO (Experimental): 30 90-minute hyperbaric oxygen sessions at 2.4 atm.
  Interventions: Procedure: Hyperbaric oxygen
- No HBO (No Intervention): No intervention. No hyperbaric oxygen is administered. Otherwise, the patient will follow the examination program.

INTERVENTIONS:
Procedure: Hyperbaric oxygen — Inhalation of 100% oxygen for 90 minutes
  Arms: HBO

SUMMARY:
Randomized clinical trial regarding the effect of hyperbaric oxygen on late radiation tissue injury to salivary gland tissue.

ELIGIBILITY:
Inclusion Criteria

* Head and neck cancer with planned radiation therapy
* Age > 18 years

Exclusion Criteria:

* Surgical treatment of head and neck cancer
* Salivary gland disease
* Severe claustrophobia
* Pregnancy or lactation (fertile women must use safe contraceptives)
* Uncontrolled hypertension (> 220/110)
* Epilepsy
* Lack of ability to equalize inner ear pressure
* Pneumothorax
* Thoracic surgery within one month before HBO treatment
* Abuse of alcohol, drugs or narcotics
* Exposed titanium surfaces or defect titanium in the oral cavity
* Previous HBO treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-05; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Salivation rate | 6 months

SECONDARY OUTCOMES:
Quality of life | 6 months
Xerostomia | 6 months
  Xerostomia questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lone Forner, DDS, PhD, Principal Investigator — Copenhagen University Hospital at Herlev
Locations (1):
- Department of Anaesthesia and Department of Oral and Maxillofacial Surgery, Copenhagen University Hospital, Copenhagen, Denmark